CLINICAL TRIAL: NCT04886648
Title: THE EFFECT OF MOTHER'S VOICE AND LULLABY ON PRETERM INFANTS' PHYSIOLOGICAL PARAMETERS, STRESS AND SLEEPING- WAKING STATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Dilek Deri̇nce Eryuruk, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Eryuruk
Record Dates: First submitted 2021-04-05; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Preterm Birth
Keywords: Mother's voice; lullaby; preterm newborn; stress; sleep-wakefulness state
MeSH Terms: conditions — Premature Birth | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: The study will be conducted in a randomized controlled manner.
Who Masked: Participant, Outcomes Assessor
Masking Description: Video footage in the study was made by three experts. Experts blindly evaluated the groups to which the videos they evaluated belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mother Voıce (Experimental): Premature baby group with mother voıce application.
  Interventions: Behavioral: Music Therapy
- Lullably (Experimental): Premature baby group with lullably application.
  Interventions: Behavioral: Music Therapy
- Control (No Intervention): Premature baby group with no application

INTERVENTIONS:
Behavioral: Music Therapy
  Arms: Lullably; Mother Voıce

SUMMARY:
The study was planned in a randomized controlled manner in order to evaluate the effect of mother's voice and lullaby on stress and sleep-wake situations of premature babies.

DETAILED DESCRIPTION:
Objective:This randomized controlled study was carried out to evaluate the effect of mother's voice and lullaby on preterm infants' stress and sleeping-waking states.

Study design:The study was carried out in a newborn unit in a public hospital in Turkey. In this study, 90 preterm newborn were divided into three groups equally as mother's voice (n=30), lullaby (n=30) and control groups (n=30). Data were obtained by Mother and Newborn Identification Form, Newborn Stress Evaluation Form (NSEF) and Newborn Sleepıng-Wakıng State Evaluation Form (NSWEF). On the 1st, 3rd and 5th days of the study; Newborns' NSEF and NSWEF scores at pre-, post-study and on the fifth minutes were evaluated. Data were evaluated by using descriptive statistics, homogeneity tests, chi-square, intra-class correlation coefficent, two way of analysis on repeated measures, generalized linear model, pearson correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* 32 0/6 -36 6 weeks of gestation
* Not connected to respiratory support device
* No surgical intervention
* Not receiving medical treatment other than appropriate vitamin supplements and antibiotic treatments
* Does not have a congenital or acquired malformation related to hearing,
* Can tolerate enterally given food (no NEC, digestive system and chromosomal abnormalities)
* The mother is at least a primary school graduate
* Diabetic mother without a baby • SGA and no IUGR

Exclusion Criteria:

Premature babies who do not meet the inclusion criteria.

-

Ages: 32 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2014-03-28 (Actual); Study Completion 2016-04-14 (Actual)

PRIMARY OUTCOMES:
Newborn Stress Evaluation Form (NSEF) | NSEF was measured on days 1 through 5, which had a 5-day application period.
  NSEF, there is no stress indicator '0', mild stress indicators' 1 ', moderate stress indicators' 2', and severe stress indicators'. It is scored as 3.

SECONDARY OUTCOMES:
Newborn Sleepıng-Wakıng State Evaluation Form (NSWEF) | NSWEF NSEF was measured on days 1 through 5, which had a 5-day application period.
  The evaluation of the newborn status was carried out under the main headings of sleep and waking behaviors. Sleep behavior; deep sleep, light sleep and drowsy. Waking behavior is grouped under the headings of awake (extremely awake and eyelids awake), active awake and crying. As a result of the evaluation, it was decided that the behaviors of the newborn were in an organized or disorganized range, and the form was marked and scoring was created for the conditions starting from the deep sleep state to disorganized crying. In the evaluation of the data; The interpretation was made according to the state score of the newborn. It was interpreted that as the YUUDF score decreased, the sleep state of the newborns increased, and as the YUUDF score increased, the wakefulness and crying status of the newborns increased.

OTHER OUTCOMES:
Heart Rate | Heart rate was measured on days 1 through 5, which had a 5-day application period.
  During the study heart rate was recorded with the help of a pulsioxymeter.
Respiratory Rate | Respiratory rate was measured on days 1 through 5, which had a 5-day application period.
  During the study, the number of respiration of preterm newborns was counted.
Oxygen Saturation | Oxygen saturation was measured on days 1 through 5, which had a 5-day application period.
  During the study, oxygen saturation was recorded with the help of a pulsioxymeter.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK ERYÜRÜK, Principal Investigator — Study Principal Investigator

IPD SHARING:
Plan to Share IPD: No
Personal data will not be shared because it was promised in the study when consent was obtained from the participants.

REFERENCES:
- [Result] Robertson AM, Detmer MR. The Effects of Contingent Lullaby Music on Parent-Infant Interaction and Amount of Infant Crying in the First Six Weeks of Life. J Pediatr Nurs. 2019 May-Jun;46:33-38. doi: 10.1016/j.pedn.2019.02.025. Epub 2019 Feb 28. PMID 30826725
- [Result] Peng NH, Chen LL, Li TC, Smith M, Chang YS, Huang LC. The effect of positioning on preterm infants' sleep-wake states and stress behaviours during exposure to environmental stressors. J Child Health Care. 2014 Dec;18(4):314-25. doi: 10.1177/1367493513496665. Epub 2013 Oct 3. PMID 24092866
- [Result] Liaw JJ, Yang L, Lee CM, Fan HC, Chang YC, Cheng LP. Effects of combined use of non-nutritive sucking, oral sucrose, and facilitated tucking on infant behavioural states across heel-stick procedures: a prospective, randomised controlled trial. Int J Nurs Stud. 2013 Jul;50(7):883-94. doi: 10.1016/j.ijnurstu.2012.08.021. Epub 2012 Oct 12. PMID 23068310
- [Result] Alipour Z, Eskandari N, Ahmari Tehran H, Eshagh Hossaini SK, Sangi S. Effects of music on physiological and behavioral responses of premature infants: a randomized controlled trial. Complement Ther Clin Pract. 2013 Aug;19(3):128-32. doi: 10.1016/j.ctcp.2013.02.007. Epub 2013 May 9. PMID 23890458
- [Result] Keith DR, Russell K, Weaver BS. The effects of music listening on inconsolable crying in premature infants. J Music Ther. 2009 Fall;46(3):191-203. doi: 10.1093/jmt/46.3.191. PMID 19757875